CLINICAL TRIAL: NCT01575938
Title: HIV Prevention Intervention for Young Transgender Women
Acronym: LifeSkills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH094323 (NIH); R01MH094323 (NIH)
Record Dates: First submitted 2012-03-29; First posted 2012-04-12 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Sexual Transmission of Infection
Keywords: HIV infection
MeSH Terms: conditions — HIV Infections | interventions — Diet; Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HIV group-based prevention intervention (Experimental): The HIV prevention intervention is a 6-session group-based and manualized intervention. Participants will also receive HIV and STI testing and counseling prior to the start of the intervention.
  Interventions: Behavioral: HIV prevention intervention
- Diet and nutrition (Active Comparator): The comparison condition is a 6-session group-based and manualized health promotion intervention. Participants will also receive HIV and STI testing and counseling prior to the start of the intervention.
  Interventions: Behavioral: Diet and Nutrition
- Standard-of-care (No Intervention): This arm will receive HIV and STI testing and counseling only.

INTERVENTIONS:
Behavioral: HIV prevention intervention — The 6-session HIV prevention intervention curriculum, "LifeSkills," incorporates interactive activities, in-depth discussions, videos, games, and role-plays to help young transgender women develop, practice, and integrate new skills into "real-life" situations. Activities address each aspect our theoretical framework (information, motivation, behavior), including experiences that may pre-dispose young transgender women to HIV/STI risk. Participants will also receive HIV and STI testing and counseling prior to the start of the intervention.
  Arms: HIV group-based prevention intervention
Behavioral: Diet and Nutrition — The comparison condition is a 6-session group-based and manualized health promotion intervention. Participants will also receive HIV and STI testing and counseling prior to the start of the intervention.
  Arms: Diet and nutrition

SUMMARY:
The purpose of this study is to test the efficacy of a uniquely targeted HIV risk reduction intervention for young transgender women (YTW), ages 16 to 29, at risk for HIV acquisition or transmission.

DETAILED DESCRIPTION:
The purpose of this study is to test the efficacy of a uniquely targeted HIV risk reduction intervention for young transgender women (YTW), ages 16 to 29, at risk for HIV acquisition or transmission. The study will test this intervention in a three-arm randomized controlled trial in two major U.S. cities with excellent access to and research experience with the population (Chicago, Boston). We will enroll at risk YTW, ages 16-29; two-fifths of the sample randomized to the intervention will participate in the 6-session group-based and manualized Life Skills intervention; two-fifths will be randomized to the standard-of-care (SOC) control condition; and one-fifth will be randomized to the time-matched attention control condition and receive standard health promotion information in a group-based multi-session format. All three arms will receive HIV and sexually transmitted infection (STI) (Chlamydia and gonorrhea) testing and pre-posttest risk reduction counseling (i.e., SOC). Sexual risk will be assessed at baseline, 4, 8 and 12 months post-randomization. Our specific aims are: 1) to determine the efficacy of the Life Skills intervention in comparison to a SOC arm and a time-matched attention control on the primary outcome: number of unprotected anal and vaginal sex acts in the previous 4 months among YTW, ages 16-29; and 2) to examine the degree to which improvements in sexual risk taking are mediated by the conceptual mediators of the intervention: transgender adaptation and integration, collective self-esteem/empowerment, information (HIV knowledge), motivation (attitudes, norms, and intentions for safer sex), and behavioral skills (discussing sex and condom use with sexual partners, acquiring and using condoms); and to explore whether reductions in sexual risk are associated with epidemiologically-linked moderators of sexual risk behavior: age, race/ethnicity, and psychosocial factors. An additional exploratory aim is to describe the prevalence of HIV and STIs in the community recruited sample; in the SOC arm, we will assess the natural trajectory of sexual risk behavior and the acquisition of HIV and STIs (incidence rate) in YTW over a 12-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* age 16-29
* self-identified as transgender, transsexual, and/or female with a male biological or birth sex
* self-reported history of unprotected anal or vaginal intercourse, anal or vaginal sex with more than one sexual partner, anal or vaginal sex in exchange for money, food, shelter, or diagnosis with HIV or another STI in the previous 4 months
* able to speak and understand English
* willing and able to provide informed consent/assent
* intention to reside in the local area throughout the 12 month follow-up period

Exclusion Criteria:

* unable to provide informed consent due to severe mental or physical illness, or substance intoxication at the time of interview
* active suicidal ideation at the time of baseline interview

Ages: 16 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in number of unprotected anal and vaginal sex acts in the previous 4 months | Baseline, 4-months post-intervention
  Self-reported unprotected anal and vaginal sex acts in the previous 4 months assessed via computer-assisted self-interviewing.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Garofalo, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Matthew Mimiaga, ScD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The Fenway Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garofalo R, Johnson AK, Kuhns LM, Cotten C, Joseph H, Margolis A. Life skills: evaluation of a theory-driven behavioral HIV prevention intervention for young transgender women. J Urban Health. 2012 Jun;89(3):419-31. doi: 10.1007/s11524-011-9638-6. PMID 22223033
- [Derived] Jin H, Restar A, Goedel WC, Ogunbajo A, Biello K, Operario D, Kuhns L, Reisner SL, Garofalo R, Mimiaga MJ. Maternal Support Is Protective Against Suicidal Ideation Among a Diverse Cohort of Young Transgender Women. LGBT Health. 2020 Oct;7(7):349-357. doi: 10.1089/lgbt.2020.0219. Epub 2020 Sep 4. PMID 32897809
- [Derived] Garofalo R, Kuhns LM, Reisner SL, Biello K, Mimiaga MJ. Efficacy of an Empowerment-Based, Group-Delivered HIV Prevention Intervention for Young Transgender Women: The Project LifeSkills Randomized Clinical Trial. JAMA Pediatr. 2018 Oct 1;172(10):916-923. doi: 10.1001/jamapediatrics.2018.1799. PMID 30105381
- [Derived] Kuhns LM, Mimiaga MJ, Reisner SL, Biello K, Garofalo R. Project LifeSkills - a randomized controlled efficacy trial of a culturally tailored, empowerment-based, and group-delivered HIV prevention intervention for young transgender women: study protocol. BMC Public Health. 2017 Sep 16;17(1):713. doi: 10.1186/s12889-017-4734-5. PMID 28915919
- [Derived] Kuhns LM, Reisner SL, Mimiaga MJ, Gayles T, Shelendich M, Garofalo R. Correlates of PrEP Indication in a Multi-Site Cohort of Young HIV-Uninfected Transgender Women. AIDS Behav. 2016 Jul;20(7):1470-7. doi: 10.1007/s10461-015-1182-z. PMID 26336946